CLINICAL TRIAL: NCT04838600
Title: A Multicenter, Prospective, Observational, Post-Market Clinical Follow-up Investigation to Confirm Clinical Performance and Safety of ChloraSolv® When Used on Chronic Leg Ulcers and Chronic Diabetic Foot Ulcers in Need of Debridement
Brief Title: A PMCF Investigation on Chronic LU and DFU in Need of Debridement With ChloraSolv®
Acronym: ChloraSolv02
Status: Terminated | Type: Observational
Why Stopped: RLS Global in bankruptcy
Sponsor: RLS Global (Industry)
Responsible Party: Sponsor
Other Study IDs: PN-00025
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-08

CONDITIONS: Chronic Leg Ulcer; Chronic Diabetic Foot Ulcer
Keywords: Leg ulcer; DFU; ChloraSolv; Debridement
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ChloraSolv — Debridement with ChloraSolv until the wound is visually assessed as clean.

SUMMARY:
This is a single-arm, observational, multicenter PMCF investigation designed to confirm clinical performance and safety of ChloraSolv when exposed to larger population of clinical users. Approximately 65 subjects will be enrolled (calculated dropout range 20%) from at least 6-12 sites in Sweden. Subjects presented with chronic leg ulcers and chronic diabetic foot ulcers in need of debridement will be enrolled and receive application of ChloraSolv per clinical routine at treating site and in accordance with the ChloraSolv Instruction for Use for up to 24 weeks. Subjects will attend a baseline visit to assess eligibility and collect demographic and baseline data and initiate treatment. There will be two follow up visits in the investigation. The first follow up visit will take place at End of Treatment, as based on investigator judgement and clinical routine at the treating site, maximum 24 weeks post baseline per the IFU. After End of Treatment, subjects will continue in the investigation with wound management per clinical routine at the treating sites for 6 weeks. At 6 weeks post End of Treatment, subjects will attend a Follow-up visit to assess safety, wound status and relative change in wound size. Besides confirmation of the clinical performance and safety when used in a larger population the investigation also includes analysis of treatment period duration. Additionally, health economy parameters will be analyzed. The investigation will be monitored to confirm the already known precautions as well as identify new precautions and possible contraindications for the use of the device. Photography of the wound pre and post debridement will be performed to confirm wound size and amount of devitalized tissue in the wound.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

1. Chronic leg ulcers and chronic diabetic foot ulcers in need of debridement
2. Male or female, 18 years of age and above
3. Able to read and understand the Patient Informed Consent and to provide meaningful written informed consent

Exclusion Criteria:

1. Known allergy/hypersensitivity to any of the components of ChloraSolv
2. Renal insufficiency defined as serum creatinine >200 μmol/L
3. Macroangiopathy expected to demand vascular intervention or percutaneous angioplasty performed less than 3 months after start of treatment; toe pressure <30mm Hg
4. Kidney or pancreas transplanted
5. Patient under cortisone treatment >60mg/day
6. Patient treated with chemotherapy or any other immune-inhibiting drugs 12 months before start of treatment
7. Other identified on-going pathologies in the area of wound, such as cancer
8. Pregnancy or breastfeeding
9. Subjects included in other ongoing clinical investigations which could interfere with this investigation, as judged by the investigator
10. Subjects not suitable for the investigation according to the investigator's judgment or other significant medical conditions that the investigator determines could interfere with compliance or investigation assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigation population will comprise of 65 subjects fulfilling the eligibility criteria of the PMCF investigation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of clean wound bed at End of Treatment, as assessed by investigator | 1 - 24 weeks
  When the investigator judges that the wound is clean primary endpoint is reached and confirmed by planimetry.

SECONDARY OUTCOMES:
Relative change in devitalized tissue and wound size at End of Treatment, compared to Baseline, assessed by planimetry | 1 - 24 weeks
  Assessed by planimetry

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jönsson, MD, Principal Investigator — Orthopedic Clinic Mölndal Hospital Sweden
Locations (7):
- Sweden (7):
  - Vårdcentralen Tunafors, Eskilstuna
  - Capio Lundby Sjukhus, Gothenburg
  - Carlanderska Hospital, Gothenburg
  - Wästerläkarna, Gothenburg
  - Wetterhälsan Munksjöstaden, Jönköping
  - Orthopedic Clinic Mölndal Hospital, Mölndal
  - Framtidens vårdavdelning, Trelleborg

IPD SHARING:
Plan to Share IPD: No
This is an observational study required by the notified body to confirm clinical performance and safety.